CLINICAL TRIAL: NCT05384938
Title: A Postmarketing, Phase 4, Multicentre, Prospective, Single-arm Study to Assess the Safety of Fasenra® (Benralizumab) in Adult Patients of Severe Asthma With Eosinophilic Phenotype in India.
Brief Title: FAsenra Safety Trial in India
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00093
Record Dates: First submitted 2021-11-09; First posted 2022-05-20 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: In Adult Patients of Severe Asthma With Eosinophilic Phenotype in India
MeSH Terms: interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, multicentre, interventional, Phase 4 study investigating the safety, tolerability, and effectiveness of Fasenra (benralizumab) in adult patients of severe asthma with eosinophilic phenotype over a period of 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benralizumab (Other): Single arm, Phase-IV
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Prospective, Single-arm Study to Assess the Safety of Fasenra® (Benralizumab) in Adult Patients of Severe Asthma with Eosinophilic Phenotype in India

SUMMARY:
Benralizumab is a humanised, afucosylated, monoclonal antibody that binds specifically to the human interlukin-5 (IL-5) receptor alpha subunit (IL-5Rα) of target cells such as eosinophils and basophils (Takatsu et al, 1994; Toba et al, 1999; Pelaia et al, 2020).

Benralizumab was generally well tolerated by patients in clinical trials, with no apparent safety concerns.

This study shall be conducted at 10 centers across India. The primary outcome measures will be

* Percentage of AEs a, SAEs, and TEAEs
* Nature, incidence, and severity of AEs including unexpected adverse drug reactions
* Percentage of patients with AEs that lead to study treatment discontinuations.

DETAILED DESCRIPTION:
Fasenra (benralizumab) has been recently approved in India with the condition to conduct a Phase 4 postmarketing study in the Indian population, as previous studies did not include patients from India. This prospective postmarketing safety study is planned to meet the regulatory mandate and assess the safety of benralizumab treatment in adult patients of severe asthma with eosinophilic phenotype over a period of 24 weeks. This interventional study will provide insights into the potential risks of eosinophil-lowering therapies when used in routine clinical care in India. The study will also evaluate the effectiveness of benralizumab in reducing asthma exacerbations.

This is a prospective, single-arm, multicentre, interventional, Phase 4 study investigating the safety, tolerability, and effectiveness of Fasenra (benralizumab) in adult patients of severe asthma with eosinophilic phenotype over a period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 75 years of age inclusive, at the time of signing the informed consent
2. Patients with physician's confirmed diagnosis of severe asthma with an eosinophilic phenotype, ie, a diagnosis of severe asthma in preceding at least 12 months, with an eosinophil count of ≥300 cells/μL at screening, requiring treatment with high-dose ICS (>500 μg fluticasone propionate dry powder formulation, or >800 μg budesonide dry powder formulation, or equivalent total daily dose) and a LABA as maintenance treatment for at least 3 months prior to enrolment
3. A decreased lung function with prebronchodilator (Pre-BD) forced expiratory volume in 1 second (FEV1) of <80% predicted, demonstrated by spirometry at screening
4. At least 2 documented asthma exacerbations in the preceeding12 months, except in 30 days before the date of informed consent, that required the use of a systemic corticosteroid or temporary increase from the patient's usual maintenance dose of oral corticosteroid (OCS)
5. Documented postbronchodilator (post-BD) reversibility in FEV1 of ≥12% and ≥200 mL in FEV1 within 12 months before first dose. If historical documentation is not available, reversibility must be demonstrated and documented at screening or Day 1 before first dose
6. Benralizumab naïve patients who have not previously received benralizumab prior to the start of this study
7. Patients who are willing and capable of giving signed informed consent as described in Appendix A, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Clinically important pulmonary disease other than asthma (eg, active lung infection, chronic obstructive pulmonary disease, bronchiectasis, pulmonary fibrosis, cystic fibrosis etc.) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome), which can confound the outcome assessment.
2. Patients currently enrolled in an interventional clinical study in parallel including those with any biologic treatment
3. Patients who have received any biologic within 30 days prior to the date of informed consent.
4. Known history of allergy or reaction to the benralizumab formulation or excipients (L-histidine, L-histidine hydrochloride monohydrate, α-trehalose dihydrate, polysorbate 20, water for injection)
5. History of anaphylaxis to any biologic therapy
6. A helminth parasitic infection diagnosed within 24 weeks before the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy
7. Acute asthma exacerbation 30 days before the date informed consent
8. Acute asthma exacerbation between screening and first dose of study dose administration.
9. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days before the date informed consent
10. Patients with malignancy within 5 years prior to enrolment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal, or squamous cell carcinoma or non-melanomatous skin cancer with active or recent malignancy
11. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis, which, in the opinion of the investigator, may put the participant at risk because of his/her participation in the study
12. History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the participant's full participation in the study, in the opinion of the investigator
13. Female patients who are pregnant or lactating or planning a family during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - Research Site, Bengaluru
  - Research Site, Chennai
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Jodhpur
  - Research Site, Lucknow
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Noida
  - Research Site, Visakhapatnam

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00093&attachmentIdentifier=6e2d1787-ecfe-4bae-b92b-32f2524e8cd6&fileName=CSR_Synopsis_FASENRA-no-proposed-redactions.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Benralizumab: 30 mg/mL subcutaneous benralizumab once every 4 weeks for the first 3 doses, followed by a maintenance dosage of 30 mg/mL once every 8 weeks thereafter
Period: Overall Study
Arm/Group | Benralizumab
Started | 139
Completed | 124
Not Completed | 15
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 6
Not completed — One participant included in study but not included in analysis as did not meet eligibility criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 67
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN | 138
  OTHER | 0
Female, Indicate childbearing potential [Count of Participants; unit: Participants] — Population: Only female participants were analyzed
  Participants
    Premenarchal: number analyzed (Participants) | 71
    Premenarchal | 0
    Premenopausal female: number analyzed (Participants) | 71
    Premenopausal female | 6
    Postmenopausal female: number analyzed (Participants) | 71
    Postmenopausal female | 30
    Potentially able to bear children: number analyzed (Participants) | 71
    Potentially able to bear children | 35

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs), Serious AEs, and Treatment-emergent AEs
Description: The number and percentage of participants who experienced at least one adverse event (AE), serious AE, or treatment-emergent AE experienced are presented
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
Participants
  Participants with at least one AE (including SAEs) | 44
  Participants with at least one serious AE | 5
  Participants with at least one treatment-emergent AE (including SAEs) | 43
  Participants with at least one non-treatment-emergent and non-serious AE | 1

2. Primary Outcome: Severity of AEs
Description: Severity of adverse events (AEs) by intensity grade
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
Participants
  Participants with at least one mild AE | 33
  Participants with at least one moderate AE | 16
  Participants with at least one severe AE | 1

3. Primary Outcome: Participants With AEs That Led to Study Treatment Discontinuations or Modifications
Description: Participants with adverse events (AEs) that led to study treatment discontinuations or modifications
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
Participants | 0

4. Secondary Outcome: Time to First Asthma Exacerbation
Description: Time to first asthma exacerbation in days in participants with asthma exacerbation
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Evaluable Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benralizumab
Number analyzed (Participants) | 19
days | 112.6 (50.45)
Statistical Analysis 1: Comparison: Benralizumab; Estimate for Time to Response (Days); Test type: Other — Single group; Median time to response = 100.0, 95% CI 2-sided [65.00 to 160.0] — Estimate for Time to Response using Kaplan-Meier method

5. Secondary Outcome: Exacerbation Rate: Before and After Treatment
Description: The annual exacerbation rate for each participant was calculated by dividing the total number of exacerbations by the number of days participated in the study and multiplying by 365.
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Evaluable Analysis Set
Measure: Mean (Standard Deviation); unit: exacerbations events/year
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
exacerbations events/year
  Exacerbation before study | 2.0 (0.00)
  Exacerbation at end of study | 0.2 (0.47)

6. Secondary Outcome: Annualized Exacerbation Rate: Overall
Description: Overall annualized exacerbation rate. The annual exacerbation rate for each participant was calculated by dividing the total number of exacerbations by the number of days participated in the study and multiplying by 365.
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Evaluable Analysis Set
Measure: Number; unit: exacerbation events/year
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
exacerbation events/year | 0.36

7. Secondary Outcome: Overall Investigators Assessment
Description: Overall investigator's assessment on the outcome of the treatment: "well controlled", "partly controlled", and "uncontrolled."
Time Frame: From study treatment to follow-up (up to 24 weeks)
Population: Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab
Number analyzed (Participants) | 135
Participants
  Well controlled | 83 [52.72 to 69.72]
  Partly controlled | 45 [25.46 to 41.96]
  Uncontrolled | 7 [2.11 to 10.39]

8. Secondary Outcome: Change in Blood Eosinophil Levels From Baseline at Weeks 4, 16, and 24
Description: Mean change in blood eosinophil levels from baseline at Weeks 4, 16, and 24
Time Frame: Baseline and Weeks 4, 16, and 24
Population: Evaluable Analysis Set
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Benralizumab
Number analyzed (Participants) | 138
cells/mm^3
  Week 4 (Visit 2) | -511 (779.13)
  Week 16 (Visit 4): number analyzed (Participants) | 133
  Week 16 (Visit 4) | -546 (867.79)
  Week 24 (Visit 5): number analyzed (Participants) | 124
  Week 24 (Visit 5) | -541 (893.62)
Statistical Analysis 1: Comparison: Benralizumab; Week 4 (Visit 2); Test type: Other — Parametric Test; p < 0.0001, paired t-test
Statistical Analysis 2: Comparison: Benralizumab; Week 16 (Visit 4); Test type: Other — Parametric Test; p < 0.0001, paired t-test
Statistical Analysis 3: Comparison: Benralizumab; Week 24 (Visit 5); Test type: Other — Parametric Test; p < 0.0001, paired t-test

ADVERSE EVENTS:
Time Frame: From screening to follow-up (up to 27 weeks)
Description: Adverse events were reported by the participant (or when appropriate by a caregiver, surrogate, or the participant's legally authorised representative). Participants were provided a patient diary to record any undesirable health-related experience or adverse events occurring during the study. Adverse events and serious adverse events mentioned both in the patient diary and verbally communicated by the participant were recorded.
Arm/Group | Benralizumab
All-Cause Mortality (participants affected / at risk) | 0/138
Serious Adverse Events (participants affected / at risk) | 5/138
Other Adverse Events (participants affected / at risk) | 39/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=138)
H1n1 influenza (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pyrexia (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=138)
Ulcer (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Sars-cov-2 test positive (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 20 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT05384938/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05384938/SAP_001.pdf